CLINICAL TRIAL: NCT04016688
Title: Comparative Study Between the Analgesic Effect of Erector Spinae Plane Block and Transversus Abdominis Plane Block After Elective Cesarean Section
Brief Title: Bilateral Erector Spinae Plane Block After Elective Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, Anesthesia lecturer, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R 126
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ES Erector Spinae Plane Block (Active Comparator): bilateral ESP block at the level of T9 by a linear ultrasound (US) transducer (Phillips Saronno Italy) placed vertically 3cm lateral to the midline to visualize the back muscles superior to the transverse process.
  A 22-G short bevel needle (spinocan, B.Braun, melsungen AG, Germany) will be inserted in cranial-caudal direction until it make contact with the transverse process. Confirmation of the correct position of the tip of the needle is by injection of 1 ml saline causing hydrodisscetion between the erector spinae muscle and the transverse process. After careful aspiration to exclude vascular puncture, 20 ml 0.25 % bupivacaine is injected.The same procedure is done on the other side of the back.
  Interventions: Procedure: ESPB and TAP block
- TAP Transversus Abdominis Plane Block (Active Comparator): bilateral TAP block: while the patient in the supine position, a linear ultrasound (US) transducer (Phillips Saronno Italy) is placed transversally on the anterolateral abdominal wall in the midaxillary line between the iliac crest and the costal margin identifying external oblique, internal oblique and transversus abdominis muscles. The TAP is between internal oblique and transversus abdominis.
  A 22-G needle (spinocan, B.Braun, melsungen AG, Germany) is introduced anteriorly to the transducer and advanced to reach the TAP between internal oblique muscle and transversus abdominis muscle. After careful aspiration to exclude vascular puncture, 20 ml 0.25 % bupivacaine is injected causing an elliptical separation of the two muscles. The same procedure is done on the other side.
  Interventions: Procedure: ESPB and TAP block

INTERVENTIONS:
Procedure: ESPB and TAP block — bilateral TAP block: while the patient in the supine position, a linear ultrasound (US) transducer (Phillips Saronno Italy) is placed transversally on the anterolateral abdominal wall in the midaxillary line between the iliac crest and the costal margin identifying external oblique, internal oblique and transversus abdominis muscles. The TAP is between internal oblique and transversus abdominis.
  A 22-G needle (spinocan, B.Braun, melsungen AG, Germany) is introduced anteriorly to the transducer and advanced to reach the TAP between internal oblique muscle and transversus abdominis muscle. After careful aspiration to exclude vascular puncture, 20 ml 0.5 % bupivacaine is injected causing an elliptical separation of the two muscles. The same procedure is done on the other side.

SUMMARY:
The aim of work is to assess and compare the analgesic efficacy of bilateral erector spinae plane block with that of bilateral transversus abdominis plane block after elective cesarean section.

DETAILED DESCRIPTION:
Inclusion criteria:

- Parturients aged 18 - 40 years with American Society of Anesthesiologists physical status І or ІІ, scheduled for elective cesarean section via a low transverse abdominal incision (Pfannenstiel) and receiving intrathecal anesthesia without sedation.

Exclusion criteria:

* Patient refusal.
* Contraindications to regional anesthesia.
* Known allergy to the study drugs.
* Severe cardiovascular, renal or hepatic diseases.
* Bleeding disorders.
* Local infection.

Participants will be randomly divided into two groups:

Group A will receive bilateral Erector spinae plane block. (n=30) Group B will receive bilateral Transversus abdominis plane block. (n=30) Simple randomization will be performed by computer-generated random numbers that will be placed in separate opaque envelopes that will be opened by responsible anesthesiologist just before the intrathecal block.

Routine preoperative investigations including electrocardiogram (ECG), complete blood picture, renal function tests, liver function tests, and coagulation profile will be done. All parturients will fast for 8 h preoperatively. IV access will be obtained (one peripheral venous cannula 18G) and standard monitoring including pulse oximetry, ECG and noninvasive blood pressure will be placed for measurement of the hemodynamic variability.

Ten ml.kg-1 of Ringer lactate solution will be infused over 15 minutes as a preload. The parturient will be asked to turn into sitting position where the skin on the back will be sterilized and spinal anesthesia will be performed via a midline approach into the L4-5 interspaces using a 25 gauge Quincke spinal needle after giving 3 ml of lidocaine 2% as a subcutaneous infiltration. After confirming free CSF flow through the needle, a 10mg of hyperbaric bupivacaine 0.5 % will be slowly injected for both groups.

The parturient will be placed in the supine position with 15° left tilt, and an oxygen mask will be applied at 2 L.min-1. The surgical procedure will start after sufficient anesthesia level is obtained, with continuous hemodynamics monitoring and recording.

After delivery of the fetus, 10 units of oxytocin will be given by IV infusion. By the end of the surgery, patients in group (A) received bilateral ESP block. First in the supine position, sham TAP block was done then the patient was turned into the lateral position to receive ESP block and after

proper skin sterilization then the vertebrae were counted from cephalad to caudal direction until T9 spinous process was reached as the first palpable spinous process is C7 and at this level a linear ultrasound (US) transducer (Phillips Saronno Italy) was placed vertically 3cm lateral to the midline to visualize the back muscles superior to the transverse process. -A 22-G short bevel needle (spinocan, B.Braun, melsungen AG, Germany) was inserted in cranial-caudal direction until it make contact with the transverse process. Confirmation of the correct position of the tip of the needle was by injection of 1 ml saline causing hydrodisscetion between the erector spinae muscle and the transverse process. After careful aspiration to exclude vascular puncture, 20 ml 0.25 % bupivacaine was injected. The same procedure was done on the other side of the back. -Patients in group (B) received bilateral TAP block. First in the supine position a linear ultrasound (US) transducer (Phillips Saronno Italy) was placed transversally on the anterolateral abdominal wall in the midaxillary line between the iliac crest and the costal margin identifying external oblique, internal oblique and transversus abdominis muscles. The TAP is between internal oblique and transversus abdominis. -A 22-G needle (spinocan, B.Braun, melsungen AG, Germany) was introduced anteriorly to the transducer and advanced to reach the TAP between internal oblique muscle and transversus abdominis muscle. After careful aspiration to exclude vascular puncture, 20 ml 0.25 % bupivacaine was injected causing an elliptical separation of the two muscles. The same procedure was done on the other side. Then the patient was placed in the lateral position to do sham ESP block.

The patients will be instructed to notify us if they have experienced any signs of systemic toxicity as circumoral or tongue numbness, dizziness, visual and auditory disturbances as difficulty focusing and tinnitus.

Spinal level will be assessed and recorded before both blocks in all patients, then they will be transferred to postoperative anesthesia care unit (PACU) with standard monitoring.

After surgery the patient will receive paracetamol 1gm IV infusion/8 hours, ketorolac 30 mg IV/12hours as a multimodal analgesia for postoperative pain.

Postoperative pain will be assessed by Visual analog scale (VAS) for pain (ranging from 0 to 10, where 0 no pain and 10 the worst possible pain) at time intervals at 0 hour, 4hours, 8 hours, 12hours and 24 hours. Postoperative mean arterial blood pressure and heart rate will be assessed and recorded.

Time for the first request to analgesia and total analgesic consumption will be recorded in the first 24 hours after surgery. Any complications as nausea and vomiting will be recorded.

Sensory block by a pin prick test will be assessed (0: normal sensation, 1: decreased pain sensation, 2: loss of pain sensation). The duration of the sensory block which is the time interval between performance of the block and complete resolution of anesthesia will be assessed and recorded every 2 hours.

Patient satisfaction with analgesia will be assessed as (0: poor, 1: good, 2: excellent).

ELIGIBILITY:
Inclusion Criteria:

* aged 18 - 40 years
* American Society of Anesthesiologists physical status ІІ, scheduled for elective cesarean section via a low transverse abdominal incision (Pfannenstiel) and receiving intrathecal anesthesia without sedation.

Exclusion Criteria:

* Patient refusal.
* Contraindications to regional anesthesia.
* Known allergy to the study drugs.
* Severe cardiovascular, renal or hepatic diseases.
* Bleeding disorders.
* Local infection.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 18 years
Enrollment: 60 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
duration of analgesia of the two blocks | 24 hours
  time

SECONDARY OUTCOMES:
Visual analogue scale | immediatiy in pacu
  Visual analogue scale for pain
Visual analogue scale | 4 hours
  Visual analogue scale for pain
Visual analogue scale | 8 hours
  Visual analogue scale for pain
Visual analogue scale | 12 hours
  Visual analogue scale for pain
Visual analogue scale | 24 hours
  Visual analogue scale for pain
the first request to analgesia | 24 hours
  duration
total analgesic consumption | 24 hours
  amount

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Faculty of Medicine, Al Fayyum
  - Mohamed Hamed, Al Fayyum
  - Mohamed, Al Fayyum

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ueshima H, Otake H. Similarities Between the Retrolaminar and Erector Spinae Plane Blocks. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):123-124. doi: 10.1097/AAP.0000000000000526. No abstract available. PMID 27997492
- [Result] Leung AY. Postoperative pain management in obstetric anesthesia--new challenges and solutions. J Clin Anesth. 2004 Feb;16(1):57-65. doi: 10.1016/j.jclinane.2003.02.012. PMID 14984863